CLINICAL TRIAL: NCT03724305
Title: Reduce Emotional Symptoms of Insomnia With Sleep Treatment
Brief Title: Reduce Emotional Symptoms of Insomnia With SleepTreatment
Acronym: RESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Christopher Drake, Principal Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESIST
Record Dates: First submitted 2018-10-25; First posted 2018-10-30 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Insomnia; Rumination
Keywords: insomnia; nocturnal rumination; depression; mindfulness; mindfulness-based therapy for insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Rumination Syndrome; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBTI (Experimental): Mindfulness-Based Therapy for Insomnia
  Interventions: Behavioral: Mindfulness-Based Therapy for Insomnia

INTERVENTIONS:
Behavioral: Mindfulness-Based Therapy for Insomnia — Mindfulness-based therapy for insomnia (MBTI) will use mindfulness-based stress reduction techniques to specifically target cognitive-emotional arousal associated with non-refractory insomnia.
  Other Names: MBTI

SUMMARY:
The purpose of this research is to test whether Mindfulness-Based Therapy for Insomnia (MBTI) significantly reduces symptoms of insomnia and cognitive arousal in patients with treatment-resistant insomnia.

DETAILED DESCRIPTION:
Cognitive-behavioral therapy and pharmacotherapy are effective interventions for insomnia. Even so, about half of patients do not adequately respond to these treatments. Non-remission has been linked to high cognitive arousal that does not improve with traditional therapies. This study will examine the effects of mindfulness-based therapy for insomnia (MBTI) in a sample of patients who previously failed cognitive behavioral therapy and/or pharmacotherapy for insomnia.

This trial utilizes a single-arm, open label trial of MBTI. MBTI is delivered via telemedicine video in an individual therapy format.

Male and female participants who have insomnia, are age 18 and older, and who are recruited into the study will complete an initial assessment of their qualifications that are based on the severity of their insomnia symptoms, depression symptoms, and physical and mental health status. Eligible participants will undergo a clinical sleep interview and then complete 8 sessions of MBTI. Study outcomes are assessed via online survey before treatment, after treatment, and then a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Determination of insomnia (ISI>10)
* Inadequate response to prior insomnia psychotherapy (e.g., CBTI) and/or pharmacotherapy per patient report.

Exclusion Criteria:

* Age < 18
* Current use of antidepressants for depression
* Bipolar or Seizure disorders
* Known sleep disorders other than insomnia (e.g. obstructive sleep apnea, narcolepsy, restless leg syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Drake, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System - Columbus, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalmbach DA, Cheng P, Ong JC, Reffi AN, Fresco DM, Fellman-Couture C, Ruprich MK, Sultan Z, Sagong C, Drake CL. Mindfulness-based therapy for insomnia alleviates insomnia, depression, and cognitive arousal in treatment-resistant insomnia: A single-arm telemedicine trial. Front Sleep. 2023 Mar 8;2:1072752. doi: 10.3389/frsle.2023.1072752. eCollection 2023. PMID 41426462

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MBTI
Started | 21
Completed | 19
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Patients with clinically significant insomnia symptoms (Insomnia Severity Index ≥ 11) and inadequate response to prior insomnia intervention per patient report.
Arm/Group | MBTI
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.16 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 12
  Race/Ethnicity: Non-Hispanic Black | 7
  Race/Ethnicity: Others | 2
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Insomnia Severity Index (ISI) Scale is a self-report measure of insomnia symptom severity. Range is 0 to 28, high score indicating a greater insomnia severity.
  units on a scale | 16.42 (3.95)
Five Facet Mindfulness Questionnaire-15 (FFMQ-15) [Mean (Standard Deviation); unit: units on a scale] — Five Facet Mindfulness Questionnaire-15 measures everyday levels of mindfulness. Scale ranges from 15 to 75 with higher scores indicating a greater level of mindfulness.
  units on a scale | 52.95 (8.30)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index
Description: Insomnia Severity Index Score (ISI; total score range 0-28, with higher scores indicating greater severity of insomnia symptoms)
Time Frame: Pre-treatment, post-treatment (7 weeks following initiation of treatment), and 6 months follow-up (6 months following conclusion of treatment)
Population: Those with clinically significant insomnia symptoms (Insomnia Severity Index ≥ 11) and inadequate response to prior insomnia intervention per patient report.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBTI
Number analyzed (Participants) | 21
score on a scale
  Pre-treatment | 16.42 (3.95)
  Post-treatment (7 weeks following initiation of treatment) | 8.37 (4.19)
  6 months follow-up (6 months following completion of treatment) | 11.72 (4.95)

2. Primary Outcome: Five Facet Mindfulness Questionnaire-15 (FFMQ-15)
Description: Five Facet Mindfulness Questionnaire - 15 (total scores ranges 15-75, with higher scores indicating someone who is more mindful in their everyday life.)
Time Frame: Pre-treatment, post-treatment (7 weeks after initiation of treatment), and 6 months follow-up (6 months following treatment conclusion)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBTI
Number analyzed (Participants) | 21
score on a scale
  Pre-treatment | 52.95 (8.3)
  Post-treatment | 57.42 (9.87)
  6 months follow-up | 55.50 (10.29)

ADVERSE EVENTS:
Time Frame: Subjects' self-report during treatment, post-treatment (7 weeks following initiation of treatment), and 6 months follow-up (6 months following conclusion of treatment)
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, doesn't differ from the clinical trials.gov definitions.
Arm/Group | MBTI
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03724305/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT03724305/ICF_001.pdf